CLINICAL TRIAL: NCT00324909
Title: Effects of Hyperbaric Oxygen Therapy on Clinical Symptoms and Markers of Inflammation and Oxidative Stress in Autistic Children: A Pilot Study
Brief Title: Effects of Hyperbaric Oxygen Therapy in Autistic Children: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hyperbarics Association (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBA-1
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2007-04-10 (Estimated); Status verified 2007-04

CONDITIONS: Autism; Oxidative Stress; Inflammation
MeSH Terms: conditions — Autistic Disorder; Inflammation | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Drug: Hyperbaric Oxygen Therapy

SUMMARY:
Autism is a neurodevelopmental disorder that currently affects as many as 1 out of 166 children in the United States. Autism is considered by many to be a permanent condition with little hope for improvement. Treatment for autism is centered on special schooling and behavioral therapy; medical science currently has little to offer.

Recent research has discovered that some autistic individuals have decreased blood flow to the brain, evidence of inflammation in the brain, and increased markers of oxidative stress. Multiple independent single photon emission computed tomography (SPECT) and positron emission tomography (PET) research studies have revealed hypoperfusion to several areas of the autistic brain, most notably the temporal regions and areas specifically related to language comprehension and auditory processing. Several studies show that diminished blood flow to these areas correlates with many of the clinical features associated with autism including repetitive, self-stimulatory and stereotypical behaviors, and impairments in communication, sensory perception, and social interaction. Hyperbaric oxygen therapy (HBOT) has been used with clinical success in several cerebral hypoperfusion syndromes including cerebral palsy, fetal alcohol syndrome, closed head injury, and stroke. HBOT can compensate for decreased blood flow by increasing the oxygen content of plasma and body tissues and can even normalize oxygen levels in ischemic tissue. In addition, animal studies have shown that HBOT has potent anti-inflammatory effects and reduces oxidative stress. Furthermore, recent evidence demonstrates that HBOT mobilizes stem cells from human bone marrow which may aid recovery in neurodegenerative diseases. Based upon these findings, it is hypothesized that HBOT will improve symptoms in autistic individuals.

The purpose of this study is to determine if HBOT improves clinical outcomes in children with autism. The study will also determine if HBOT changes markers of inflammation and oxidative stress in autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with autism spectrum disorder

Exclusion Criteria:

* Seizures not controlled by medicine
* Inability to ventilate ears

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 18

PRIMARY OUTCOMES:
Scores on autism rating scales before and after HBOT
Measure of inflammation before and after HBOT
Measures of oxidative stress before and after HBOT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Rossignol, MD, Principal Investigator — Blue Ridge Medical Center
Locations (1):
- Blue Ridge Medical Center, Arrington, Virginia, United States

REFERENCES:
- [Derived] Rossignol DA, Rossignol LW, James SJ, Melnyk S, Mumper E. The effects of hyperbaric oxygen therapy on oxidative stress, inflammation, and symptoms in children with autism: an open-label pilot study. BMC Pediatr. 2007 Nov 16;7:36. doi: 10.1186/1471-2431-7-36. PMID 18005455